CLINICAL TRIAL: NCT06009978
Title: The Effect of Early Treatment With Neuromuscular, Electrical Stimulation (NMES) After Achilles Tendon Rupture
Brief Title: Effect of Additional Treatment With NMES After Achilles Tendon Rupture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00921-02
Record Dates: First submitted 2023-07-10; First posted 2023-08-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Achilles Tendon Rupture; Physical Disability
Keywords: Achilles Tendon Rupture; Rehabilitation; Neuromuscular Electrical Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional treatment with NMES after Achilles Tendon rupture (Active Comparator): Neuromuscular electrical stimulation 2 times a day á 15 minutes during the week 3-8 after the Achilles Tendon rupture.
  Patients will also follow ordinary standard rehabilitation for Achilles Tendon rupture
  Interventions: Device: Neuromuscular electrical stimulation (NMES)
- Control group (No Intervention): Patients will follow ordinary standard rehabilitation for Achilles Tendon rupture

INTERVENTIONS:
Device: Neuromuscular electrical stimulation (NMES) — Neuromuscular electrical stimulation (NMES) 2 times a day á 15 minutes from the third to the eight week after injury. The additional treatment will be perform in the patients home by themselves
  Arms: Additional treatment with NMES after Achilles Tendon rupture

SUMMARY:
Increased knowledge is needed about new methods how to treat patients with Achilles tendon ruptures (ATR). A goal is to be able to individualize as well as improve treatment beyond the question about if surgery should be used or not.

An overall aim of the project is to, in a randomized controlled trial (RCT), explore what impact a new treatment method with Neuromuscular Electrical Stimulation (NMES) - attached on the patients ́ calf muscles on the injured leg - in the early stages after an ATR, may have on tendon length, functional performance, biomechanical variables and patient reported outcome, both in the short and long term after the injury. 70 patients are planned to be included in this RCT and will be evaluated 3,6 and 12 months after their injury. Primary outcome will be heel-rise height. Secondary outcome will be tendon length, jumping ability, patient- reported outcome and biomechanical loading pattern.

There is also a need to explore if the patients ́ loading patterns improve after treatment with NMES. Therefore, biomechanical variables in lower leg during walking and jumping will also be evaluated one year after their injury.

The planned studies include completely new ways of exploring how to optimize the rehabilitation after an ATR.

Since there might be an increased risk for overuse injuries in the healthy limb, there will also be focus on how the non- injured limb may be affected of an ATR.

Taken together, this new knowledge can be helpful in the clinical setting to individualize and optimize patients' treatment and rehabilitation with the goal to guide the patient return to the same, or higher level of, physical activity as before the injury.

DETAILED DESCRIPTION:
BACKGROUND:

There is limited knowledge about how calf muscle performance and tendon elongation affect the patient's discomfort or ability to return to previous activity levels after an Achilles Tendon rupture. Tendon elongation can cause a changed recruitment pattern of the different parts of the muscle complex triceps surae. There is some evidence that treatment with Neuromuscular Electrical Stimulation (NMES) can improve postural balance by stimulating the calf muscles in elderly people with impaired balance. A newly published study concluded that NMES treatment the first 12 weeks after an ATR, did not have any impact on calf circumference or patient-reported outcome the first 12 weeks after the injury.

Studies have shown that only 20-40% of patients are able to return to the same level of physical activity as before the injury. Although patients return to full participation in sports, their level of performance is often adversely affected. Obviously, there can be different reasons for this. In a newly published study, it was concluded that joint power distribution during a drop countermovement jump was affected by fear of reinjury as long as 2 years after an ATR. However, there is still a lot to explore about if an improved physical function in the injured calf muscle may decrease the fear of re-injury and therefore positively affect the ability to return to previous physical activity level after an ATR. Therefore, new treatments with the goal to increase the possibility to return to the same physical level as before the injury are very much needed.

An ATR can lead to reduced strength development in the ankle with simultaneous increased load development in the knee joint in the injured leg for as long as 6 years after the injury. Reduction in strength and endurance in the calf muscle has been shown to persist long after the injury. Exhaustion of the lower leg muscles affects the valgus moment in the knee as well as kinematic variables in athletes during vertical jumps, which may affect the risk of knee injury. However, there is a lack of knowledge about how lower leg function, biomechanics and muscle recruitment are affected in patients after an ATR. It is also unknown how this injury affects the healthy limb and perhaps increase the risk of overload injuries in other parts of the body.

HYPOTHESIS:

Additional treatment with NMES in early stages after an Achilles Tendon rupture have a positive impact on lower leg function both in the short and long term.

PURPOSE AND SPECIFIC GOALS:

An overall aim of the project is to, in a randomized controlled trial, explore what impact a new treatment method with NMES in the early stages after an ATR may have on calf muscle performance, tendon length, jumping ability, biomechanical variables and patient reported outcome both in the short and long term after the injury.

There will also be focus on how the non-injured limb may be affected of an Achilles tendon rupture. This new knowledge can be helpful in the clinical setting to

1. individualize and optimize patients' treatment and rehabilitation
2. avoid overuse injuries, both in the injured and healthy limb The goal will be to guide the patient return to the same, or higher level of physical activity as before the injury.

OBJECTIVES:

* To explore if additional treatment with NMES during the first 3-8 weeks after an ATR can improve calf muscle function, biomechanical variables, tendon lengthening and patient-reported outcome both in short an long term. The design of this study is a Randomized Controlled Trial (RCT).
* To evaluate the biomechanics of the ankle, knee and hip during walking, running and jumping in both limbs in two groups of patients one year after an ATR. One group has been treated with NMES 3-8 weeks after the injury and the other group has not.

METHOD The design of this study is a randomized controlled trial. A power calculation (p <0.05, power 80%) showed that 28 patients who receive and 28 who do not receive treatment with NMES are needed to be able to show a clinically important difference of 10% in heel-rise height. A total of 70 patients with ATR will be included and randomized to receive or to not receive additional therapy with NMES during the first 3-8 weeks after their ATR.

Four electrodes connected with the NMES equipment will be attached on the patients ́ calf on the injured leg and they will use the equipment in their home two times a day á 15 minutes for six weeks, that is 3-8 weeks after the injury.

Primary outcome will be the heel-rise height during the heel-rise work test. Standardized seated heel-rise as well as single-leg standing heel- rise will be evaluated 3, 6 and 12 months after the injury in both the injured and the healthy limb. The heel-rise work test will be evaluated with a linear encoder connected to the software MuscleLab®.

Tendon length will be evaluated with ultrasound 8 weeks and 3, 6 and 12 months after the injury. The measurement is found to be reliable and valid. The tendon length will be evaluated with ultrasonography with extended field of view using a wideband array linear probe (5.0- 13.0 MHz). The B- mode at 10 MHz and a depth of 3 cm will be used to record the images.

One year after the injury, kinematic and kinetic variables together with EMG will be evaluated during walking, running and jumping. For collection of the biomechanical data, 16 7+ cameras and 4 force plates will be used. This new equipment is available in a new motional analysis lab at our research unit. Fifty-five reflectors will be attached on the patients´ body to be able to detect segmental movements. EMG electrodes on the medial and lateral Gastrocnemius, Soleus and Tibialis anterior muscles will also be attached on the patient in order to measure how the muscles are recruited in the different activities. Both healthy and injured sides will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Achilles Tendon rupture
* The injury should have been treated within two days from the trauma
* The rupture is located in the mid portion of the tendon

Exclusion Criteria:

* Pregnancy
* Having a pace maker, intra cardiac defibrillator or other active implant
* Having had an Achilles Tendon rupture before, regardless of side
* Having an earlier injury that will have an impact on lower leg function, regardless of side
* Diabetes
* Neuro vascular disease
* Immunosuppressive treatment
* Difficulties to understand the language or difficulties in understand instructions.
* Unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Heel-rise height during heel-rise work test | 12 months
  Evaluation of heel-rise height during heel-rise work test. Comparison between groups in heel-rise height Limb Symmetry Index (LSI) - injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome
Heel-rise height during heel-rise work test | 6 months
  Evaluation of heel-rise height during heel-rise work test. Comparison between groups in heel-rise height (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome
Heel-rise height during heel-rise work test | 3 months
  Evaluation of heel-rise height during heel-rise work test using. Comparison between groups in heel-rise height (LSI)- injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome

SECONDARY OUTCOMES:
Tendon length | 12 months
  Comparison between groups and limbs in Length measured with ultrasound from insertion to myotendinous junction in both limbs.
Tendon length | 6 months
  Comparison between groups and limbs in Length measured with ultrasound from insertion to myotendinous junction in both limbs.
Tendon length | 3 months
  Comparison between groups and limbs in Length measured with ultrasound from insertion to myotendinous junction in both limbs.
Gastrocnemius Cross-sectional area | 12 months
  Comparison between groups and limbs in Area of medial and lateral gastrocnemius in both limbs
Gastrocnemius Cross-sectional area | 6 months
  Comparison between groups and limbs in Area of medial and lateral gastrocnemius in both limbs
Gastrocnemius Cross-sectional area | 3 months
  Comparison between groups and limbs in Area of m medial and m lateral gastrocnemius in both limbs
Soleus cross-sectional area | 12 months
  Comparison between groups and limbs in Area of m soleus in both limbs
Soleus cross-sectional area | 6 months
  Comparison between groups and limbs in Area of m soleus in both limbs
Soleus cross-sectional area | 3 months
  Comparison between groups and limbs in Area of m soleus in both limbs
Biomechanical data; kinematic data will be evaluated during walking, running and jumping. | 12 months
  16 7+ cameras and 4 force plates will be used. 55 reflectors will be attached on the patients´body to be able to detect segmental movements. Kinematic data will be evaluated in degrees in ankle, knee and hip. Comparison will be performed between groups and limbs in degrees (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome.
Biomechanical data; kinetic data will be evaluated during walking, running and jumping. | 12 months
  16 7+ cameras and 4 force plates will be used. 55 reflectors will be attached on the patients´body to be able to detect segmental movements. Kinetic data will be evaluated in power (watt) in ankle, knee and hip. Comparison will be performed between groups and limbs in power (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome.
Electro Myography (EMG) will be evaluated during walking, running and jumping. | 12 months
  EMG electrodes on the medial and lateral Gastrocnemius, Soleus and Tibialis anterior, Quadriceps and trunk muscles will be attached on the patient in order to measure how the muscles are recruited during walking running and jumping. Both healthy and injured sides will be analyzed. The electrical activity in the muscles will be evaluated. Comparison will be performed between groups and limbs in power (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome.
Achilles tendon Total Rupture Score (ATRS) | 3 months
  A valid and reliable questionnaire developed for patients with an Achilles Tendon rupture with a purpose to evaluate patient reported outcome in terms of symptoms and function. The values can be between 0 and 100 and the higher score, the better outcome.
Achilles tendon Total Rupture Score (ATRS) | 6 months
  A valid and reliable questionnaire developed for patients with an Achilles Tendon rupture with a purpose to evaluate patient reported outcome in terms of symptoms and function.The values can be between 0 and 100 and the higher score, the better outcome.
Achilles tendon Total Rupture Score (ATRS) | 12 months
  A valid and reliable questionnaire developed for patients with an Achilles Tendon rupture with a purpose to evaluate patient reported outcome in terms of symptoms and function.The values can be between 0 and 100 and the higher score, the better outcome.
Physical Activity Scale (PAS) | 12 months
  A patient reported outcome used for the purpose to evaluate the patients self estimated physical activity level. The scale is from 1 to 6 and the higher score, the better outcome.
Physical Activity Scale (PAS) | 6 months
  A patient reported outcome used for the purpose to evaluate the patients self estimated physical activity level.The scale is from 1 to 6 and the higher score, the better outcome.
Physical Activity Scale (PAS) | 3 months
  A patient reported outcome used for the purpose to evaluate the patients self estimated physical activity level.The scale is from 1 to 6 and the higher score, the better outcome.
Drop Countermovement Jump | 6 months
  Drop Countermovement Jump: Evaluation of vertical jumping height after jumping from a 20 cm high box. The outcome will be measured as the height the patient can perform in jump height after landing in cm. Comparison between groups and limbs in jump height will be presented as Limb Symmetry Index (LSI)- injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Drop Countermovement Jump | 12 months
  Drop Countermovement Jump: Evaluation of vertical jumping height after jumping from a 20 cm high box. The outcome will be measured as the height the patient can perform in jump height after landing in cm. Comparison between groups and limbs in jump height will be presented as Limb Symmetry Index (LSI)- injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Hopping | 6 months
  Evaluation of series of jumps as in jumping ropes. The outcome measurement will be mean jumping height in cm and elasticity ratio in 20 jumps. Comparison between groups and limbs in jump height and elasticity ratio will be presented as Limb Symmetry Index (LSI)- injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Hopping | 12 months
  Evaluation of series of jumps as in jumping ropes. The outcome measurement will be mean jumping height in cm and elasticity ratio in 20 jumps. Comparison between groups and limbs in jump height and elasticity ratio will be presented as Limb Symmetry Index (LSI)- injured side/healthy side *100 expressed in percent. The range in LSI is between 0-100% and the higher value, the better outcome.
Calf muscle power | 6 months
  Evaluation of calf muscle power in a weight training machine expressed in watt (Newton x meter /seconds). Comparison will be performed between groups and limbs in power (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome.
Calf muscle power | 12 months
  Evaluation of calf muscle power in a weight training machine expressed in watt (Newton x meter /seconds). Comparison will be performed between groups and limbs in power (LSI)- injured side/healthy side *100 expressed in percent.The range in LSI is between 0-100% and the higher value, the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Nilsson Helander, Ass.Prof, Principal Investigator — VGregion
Locations (1):
- Forskningsenhet Ortopedi, Sahlgrenska universitetssjukhuset, Mölndal, Mölndal, VGregion, Sweden

IPD SHARING:
Plan to Share IPD: No